CLINICAL TRIAL: NCT05313776
Title: Identification of Non-motor Brain Areas Involved in Upper Limb Motor Recovery After Stroke
Acronym: NOMO-Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other); Euromov, Université Montpellier (Unknown); IMT Mines Ales (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0431
Record Dates: First submitted 2022-02-23; First posted 2022-04-06 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Upper Limb Ischemia; Stroke
Keywords: Ischemic stroke; Motor recovery; Upper-limb; Functional MRI; Neuroplasticity
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-stroke: People with a first ever ischemic stroke of the middle cerebral artery presenting severe motor deficits of the upper-limb at onset.
  The patients
  Interventions: Other: Magnetic Resonance Imaging
- Controls: Age and sexe matched healthy subjects without known neurological and or psychological deficits.
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — IMR is a non-invasive imaging technology that produces three dimensional detailed anatomical images. It is often used for disease detection, diagnosis, and treatment monitoring. It is based on sophisticated technology that excites and detects the change in the direction of the rotational axis of protons found in the water that makes up living tissues.

SUMMARY:
Why: Upper-limb recovery post-stroke is challenging. Rehabilitation, aiming to induce plasticity takes an important place in patients' treatment. The last years, non-invasive brain stimulation of the primary motor cortex has gained the communities' interest, allowing direct modification of neural excitability and thus impacting plasticity. Yet, research outcomes remain inconclusive to date. It's expected this to be related to patient heterogeneity including mild to severe motor deficits, and suboptimal site of stimulation. It might be questioned whether M1 stimulation is preferable over that of higher association areas like the parietal or premotor cortex.

What: The aim of the study is to identify alternative brain regions to stimulate, related to improved motor quality after a severe initial deficit. How: by following motor recovery over time, by co-recording movement kinematics and brain activity.

Because: Stimulation of the novel identified regions may improve motor recovery after stroke.

DETAILED DESCRIPTION:
Patients' brain activity and connectivity during an elbow flexion/extension task will be evaluated at 2 weeks (V0), 3 months (V1) and 6 months (V2) post-stroke. Between V0 and V1, patients will receive standard in-care rehabilitation at the physical and rehabilitation medicine department (PMR) of Montpellier's University Hospital: 120 minutes a day, for 5 days/week (orthopedic training, sitting/standing balance, walking, sensorimotor training - including 2 and 3 dimensional reach to grasp exercises with and without vision, functional electrical stimulation of the upper-limb, finger pinching exercises). On the day of imaging, a clinical evaluation will be performed to evaluate patients upper-limb function (Fugl-Meyer Upper Extremity scale) and capacity (WOLF motor function test & Box and Block test). The imaging protocol includes a 3DT1 for anatomical reference, a functional task-based MRI with block-design (30s rest alternated with 30s of activity) and diffusion tensor imaging (DTI) to quantify anatomical connectivity. During imaging, participants will lay on their back with their arm stretched along their body. A short auditory signal will inform patient when to start/stop moving. During movement, only the elbow will be rhythmically flexed and extended at a self-selected comfortable pace in the vertical plane. The motor task will be performed with both the paretic and ipsilesional upper-limb, in random order. Patients that are unable to move, will be asked to keep trying to move during the activity block.

Material: 3.0T whole-body magnet MRI (Prisma Siemens, Germany), MRI compatible 3D motion camera's (Qualisys, France).

Imaging data will be acquired by the I2FH research platform at the Montpellier University Hospital Data treatment: functional Imaging data will be preprocessed following standard procedures, including reorientation to the anterior commissure, slice-time correction, realignment, co-registering & normalization to 3DT1 anatomical template, smoothing. Subsequent group analyses using general linear models, will be corrected for multiple comparisons. Imaging data will be analyzed by the I2FH research platform. 3D-Movement time-series of upper-limb displacement will be analyzed by Euromov, using matlab the mathworks. The movement will be quantified by its shaping (e.g. Amplitude/Frequency) and structure (e.g. Fluency/Directness). Clinical testing will be performed as part of standard care evaluations at the physical rehabilitation medicine department of the hospital of Montpellier and Nimes.

Schedule visit:

Patients: V0: ~10 post-stroke, V1: ~3 months post-stroke, V2: ~6 months post stroke. Clinical testing will be performed on the day (+/- 1) of the MRI session.

Healthy subjects will be evaluated once

ELIGIBILITY:
Inclusion Criteria patients post-stroke:

* 18-85 yrs,
* First ever ischemic stroke of the middle cerebral artery,
* Initial severe motor deficit (fugl-Upper limb assessment score <30/66),
* Written consent.

Exclusion criteria patients post-stroke:

* The presence of secondary neurological or psychiatric deficits,
* Strong hemineglect (bell-test);
* Aphasie >3/5 on the Boston scale,
* Bilateral stroke,
* Hemorraghic stroke,
* MRI contra-indications,
* Pregnancy/breastfeading,
* Patient under curatele,
* Medical urgency.

Inclusion criteria healthy subjects:

* Age matching (+/- 5 yrs),
* Sexe matching,
* Written consent.

Exclusion criteria healthy subjets:

* Neurological or psychological deficits;
* MRI contra-indations;
* Pregnancy/breastfeeding,
* Personunder curatele.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted at the University hospital of Montpellier with an ischemic stroke that are meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change of brain activity during motor task during post-stroke recovery | ~10days, 3 months and 6 months post-stroke.
  Functional MRI imaging with upper-limb elbow flexion in a blocked-design. Analysis with integrated movement kinematics that are registered simulateously.

SECONDARY OUTCOMES:
fMRI task-based and resting state brain connectivity | at ~10days, 3 months and 6 months post-stroke.
  Resting-state and functional MRI with upper-limb elbow flexion
Diffusion Tensor Imaging anatomical brain connectivity | at ~10days, 3 months and 6 months post-stroke.
  DTI imaging

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LAFFONT, PHD,MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France